CLINICAL TRIAL: NCT02370524
Title: Quantitative Evaluation of [18F]T807 as a Potential PET Radioligand for Imaging Tau in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Molecular NeuroImaging (Other)
Collaborators: Institute for Neurodegenerative Disorders (Other); Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Danna Jennings, Principal Investigator, Molecular NeuroImaging
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: [18F]T807
Record Dates: First submitted 2015-02-17; First posted 2015-02-25 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Alzheimer's Disease (AD)
MeSH Terms: conditions — Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole; florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18F]T807 (Experimental): At the [18F]T807 PET imaging visit, subjects will be given a bolus injection of no more than 10 mCi (370 MBq) of [18F]T807
  Interventions: Drug: [18F]T807

INTERVENTIONS:
Drug: [18F]T807 — All enrolled subjects will undergo an [18F]T807 PET imaging visit. In addition, subjects with AD and aged volunteers will have one PET scan with Amyvid (florbetapir F 18 injection) as part of the screening activities to measure Aβ in the brain.
  Other Names: Amyvid; [18F]florbetapir

SUMMARY:
The primary objective of this exploratory imaging study is to further characterize [18F]T807, an investigational PET radioligand for imaging Tau (thought to be a downstream biomarker indicative of neurodegeneration in conditions such as AD).

ELIGIBILITY:
Inclusion Criteria:

For all Subjects:

* Written informed consent or assent is obtained
* Female subjects/volunteers must be either surgically sterile (by means of hysterectomy, bilateral oophorectomy, or tubal ligation) or post-menopausal for at least 1 year or, if they are of childbearing potential, must commit to the use of two effective contraception methods for the duration of the study.
* Male subjects/volunteers and their partners of childbearing potential must commit to the use of two effective methods of contraception, one of which should be a barrier method for male subjects.

Prodromal and Mild Alzheimer's Disease Subjects

* Males and females aged between 50 and 90 years.
* Study partner has noticed a recent gradual decrease in the subject's memory (e.g., over the prior 12 months), which the subject may or may not be aware of.
* For prodromal subjects, abnormal memory function at screening or 4 weeks prior to screening based on the FCSRT-IR of:Free recall <17, or Total recall <40, or Free recall <20 and total recall <42.
* Individuals with mild AD must meet the criteria based on the National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association and Diagnostic and Statistical Manual of Mental Disorders, Version 5, criteria. This evidence may be compiled during screening but must be fully documented in the subject's study file before the baseline visit.
* Have an MMSE (Folstein et al. 1975) score at screening >20.
* Have an Amyvid (florbetapir F 18 injection) scan at screening that demonstrates amyloid binding based on qualitative analysis (visual read) that meets the criteria for AD.
* Modified Hachinski Ischemia Scale (Moroney et al. 1997) score of ≤ 4.
* A neuroimaging evaluation of the brain by MRI that supports a diagnosis of AD with no evidence of focal disease to account for dementia or MRI exclusion criteria.
* Medications taken for symptomatic treatment of AD must be maintained on a stable dosage regimen for at least 4 weeks before the [18F]T807 imaging visit.
* Able to participate in all scheduled evaluations.
* The subject has an appropriate caregiver or community dwelling with a caregiver capable of accompanying the subject on all visits to the center as judged by the investigator.
* In the opinion of the investigator, the subject and caregiver will be compliant and have a high probability of completing the study.

Healthy Volunteers

* Males and females aged between 20 and 90 years. Younger healthy controls will be aged 20-49 and older healthy controls will be aged 50-90.
* Healthy volunteers with no clinically relevant findings on physical examination at screening and upon reporting for the [18F]T807 imaging visit.
* No suspicion of cognitive impairment/early dementia from MMSE as judged by the investigator (MMSE>28).
* No concomitant medications, over-the-counter, supplement, or any other agent intended to improve cognition or prevent cognitive decline
* A negative Amyvid (florbetapir F 18 injection) scan at screening based on qualitative analysis (visual read).

Exclusion Criteria:

For All subjects:

* Current or prior history of any alcohol or drug abuse.
* Severe systemic disease based on history and physical examination.
* Positive result on urine screen for illicit drugs.
* Laboratory tests with clinically significant abnormalities
* Clinically significant unstable medical or psychiatric illness.
* Positive test for hepatitis B or C or HIV.
* Prior participation in other research protocols or clinical care in the last year such that radiation exposure is >15 mSv and participation in this study would require the subject/volunteer to exceed the annual limits.
* Pregnancy or breastfeeding.
* Current or prior history of coagulopathy.
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* History of significant drug and/or food allergies, anaphylactic/anaphylactoid reaction to any allergen.
* Contraindication for arterial cannulation.
* Unsuitable veins for repeated venipuncture.
* MRI exclusion criteria include: non-AD pathology such as infectious disease, space-occupying lesions, normal pressure hydrocephalus, or any other abnormalities associated with significant CNS disease
* Any lacunar infarct in a strategically important location known to lead to cognitive impairment such as the thalamus, hippocampus of either hemisphere, or head of the left caudate
* Severe sub-cortical microvascular disease (Fazekas score of 3 for deep white matter hyperintensities) (Fazekas et al. 1987)
* Territorial infarct or macroscopic hemorrhage (>10 mm)
* Implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips or other medical implants that have not been certified for MRI, or history of claustrophobia in MRI
* Observed claustrophobia at screening
* Ferromagnetic foreign bodies, such as metal shrapnel or bullet fragments, need to be considered on an individual basis

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Quantitative evaluation of [18F]T807 as a potential PET radioligand for imaging Tau in patients with clinically characterized tauopathies | 1 year
  To further characterize [18F]T807, an investigational PET radioligand for imaging Tau (thought to be a downstream biomarker indicative of neurodegeneration in conditions such as AD) and to assess the full quantitative evaluation of the PET outcome measures using [18F]T807 by pharmacokinetic (PK) modeling in order to derive a volume of distribution (VT) of [18F]T807 using arterial input function.

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Molecular NeuroImaging, LLC, New Haven, Connecticut, United States

REFERENCES:
- [Background] Fazekas F, Chawluk JB, Alavi A, Hurtig HI, Zimmerman RA. MR signal abnormalities at 1.5 T in Alzheimer's dementia and normal aging. AJR Am J Roentgenol. 1987 Aug;149(2):351-6. doi: 10.2214/ajr.149.2.351. PMID 3496763
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Moroney JT, Bagiella E, Desmond DW, Hachinski VC, Molsa PK, Gustafson L, Brun A, Fischer P, Erkinjuntti T, Rosen W, Paik MC, Tatemichi TK. Meta-analysis of the Hachinski Ischemic Score in pathologically verified dementias. Neurology. 1997 Oct;49(4):1096-105. doi: 10.1212/wnl.49.4.1096. PMID 9339696
- [Derived] Barret O, Alagille D, Sanabria S, Comley RA, Weimer RM, Borroni E, Mintun M, Seneca N, Papin C, Morley T, Marek K, Seibyl JP, Tamagnan GD, Jennings D. Kinetic Modeling of the Tau PET Tracer 18F-AV-1451 in Human Healthy Volunteers and Alzheimer Disease Subjects. J Nucl Med. 2017 Jul;58(7):1124-1131. doi: 10.2967/jnumed.116.182881. Epub 2016 Dec 1. PMID 27908967
- See also: Molecular NeuroImaging — http://www.mnimaging.com
- See also: Institute for Neurodenerative Disorders — http://www.indd.org